CLINICAL TRIAL: NCT00705809
Title: T-Cell Project: Epidemiologic Component
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908163; 08-C-N163
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-20

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Epidemiology; Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The T-Cell Project, sponsored by the International T-cell non-Hodgkin Lymphoma Study Group, is a consortium of institutions interested in achieving more detailed information on clinical and biological characteristics of T-cell lymphomas.
* The T-Cell Project serves as a repository for data on patients with peripheral T-cell lymphoma (PTCL) worldwide. Its overall goal is to improve T-cell subtype classifications and evaluate treatment strategies for each subtype.

Objectives:

-To implement a standardized epidemiologic questionnaire into the ongoing T-Cell Project to allow evaluation of various potential risk factors for PTLCs.

Eligibility:

-Untreated patients 18 years of age and older who were diagnosed with PTLC September 1, 2006, or later.

Design:

-Patients complete a questionnaire containing the following information:

Demographic information

Smoking history and alcohol use

Personal history or cancer

History of cancer among first-degree relatives

Medical history

History of transplants

History of blood transfusions

Medication use

Occupational and residential history

Pesticide treatment

-The information collected is linked to clinical and pathologic information in the T-Cell Project database.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCLs) comprise a heterogeneous group of neoplasms that are derived from post-thymic lymphoid cells at different stages of differentiation with different morphological patterns, phenotypes, and clinical presentations. Although a number of case-control studies on non-Hodgkin lymphoma (NHL) have identified various risk factors for disease, including autoimmune conditions, family history of hematopoietic malignancies, smoking, hepatitis C infection, and host susceptibility, these risk factors largely pertain to B-cell lymphoma subtypes as they comprise well over 90 percent of all NHLs. At present, there are no known epidemiologic risk factors for PTCL or its subtypes. This is largely due to the lack of sample size of PTCL in any one epidemiologic study. The aim of this proposal is to implement a standardized epidemiologic risk factor questionnaire into the on-going T-Cell Project. Briefly, the T-Cell Project is an international consortium of on-going clinical trials on peripheral PTCL. It serves as a prospective collection of patients (greater than 18 years) worldwide with PTCL who are enrolled at participating medical institutions for treatment in a clinical trial. The overall goal of the T-Cell Project is to improve current T-cell subtype classifications and to evaluate different treatment strategies for each T-cell subtype. The specific goal of our proposal is to implement, within the T-Cell Project, a 20-minute standardized epidemiologic questionnaire to allow evaluation of various potential risk factors for T-cell lymphomas. Importantly, there are currently no known epidemiologic risk factors for PTCL. We plan to administer questionnaires to 800 PTCL patients; if successful this collection would be the largest database of PTCLs to date with epidemiologic data. If the questionnaire implementation of assessing epidemiological risk factors for PTCL among patients in the T-Cell Project is found logistically feasible, then descriptive and analytic epidemiologic analyses of the collected data to understand the etiology of PTCL would be pursued at the NCI in collaboration with members of the T-Cell Project. For such analyses, NCI would receive only fully anonymized and de-linked data with no identifiers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years
* Histologically confirmed Periperal T-cell lymphoma on or after September 1, 2006

EXCLUSION CRITERIA:

* Age less than 18 years
* Cases without histological confirmation
* Cases diagnosed prior to September 1, 2006

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-06-18; Study Completion 2011-07-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Delves PJ, Roitt IM. The immune system. Second of two parts. N Engl J Med. 2000 Jul 13;343(2):108-17. doi: 10.1056/NEJM200007133430207. No abstract available. PMID 10891520
- [Background] Delves PJ, Roitt IM. The immune system. First of two parts. N Engl J Med. 2000 Jul 6;343(1):37-49. doi: 10.1056/NEJM200007063430107. No abstract available. PMID 10882768
- [Background] Jones D, O'Hara C, Kraus MD, Perez-Atayde AR, Shahsafaei A, Wu L, Dorfman DM. Expression pattern of T-cell-associated chemokine receptors and their chemokines correlates with specific subtypes of T-cell non-Hodgkin lymphoma. Blood. 2000 Jul 15;96(2):685-90. PMID 10887135